CLINICAL TRIAL: NCT06955234
Title: Berbevis Project: Multitarget Dose-finding Study
Brief Title: Berbevis Dose-finding Study in Subjects With Impaired Fasting Glucose
Acronym: BERBEVIS-DFG-0
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508/29032024; 1508/29032024 (Other: Ethics Committee IRCCS Policlinico San Matteo)
Record Dates: First submitted 2025-04-17; First posted 2025-05-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Impaired Fasting Glucose (IFG)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Berbevis 500 mg/die (Experimental): Berbevis™, 250 mg x 2/day, 1 tablet in the morning and 1 in the evening.
  Interventions: Dietary Supplement: Berbevis supplement
- Berbevis 750 mg/die (Experimental): Berbevis™, 250 mg x 3/day, 2 tablets in the morning and 1 in the evening.
  Interventions: Dietary Supplement: Berbevis supplement
- Berbevis 1000 mg/die (Experimental): Berbevis™, 250 mg x 4/day, 2 tablets in the morning and 2 in the evening.
  Interventions: Dietary Supplement: Berbevis supplement

INTERVENTIONS:
Dietary Supplement: Berbevis supplement — This intervention consists of a standardized oral dietary supplement containing Berberis aristata extract formulated in phospholipids (Berbevis™). The supplement is formulated to support metabolic balance. It is administered twice daily for 8 weeks to evaluate safety, tolerability, and dose-response effects in healthy adult volunteers.

SUMMARY:
Assessing the effects of a nutraceutical supplement (Berbevis™) in adults with impaired fasting glucose (100-126 mg/dL) and BMI between 25 and 35. Ninety participants will be assigned to three parallel groups receiving Berbevis™ at increasing daily doses (500 mg, 750 mg, and 1000 mg) for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* fasting blood glucose between 100 and 126 mg/dl
* BMI between 25 and 35 kg/m^2

Exclusion Criteria:

* Fasting blood glucose below 100 mg/dl
* BMI < 25 or > 35 kg/m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in fasting blood glucose levels from baseline after 4 weeks of Berbevis™ supplementation | 4 weeks
  Fasting blood glucose levels will be measured at baseline and after 4 weeks of supplementation with Berbevis™ using standard blood chemistry analysis.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) during 4 weeks of Berbevis™ supplementation at different dosages | 4 weeks
  Safety will be assessed by monitoring the occurrence of AEs and SAEs during the 4-week supplementation period. Events will be recorded by investigators and reported according to current GCP and pharmacovigilance regulations.
Change from baseline in lipid profile (total cholesterol, HDL, LDL, Apo A, Apo B, triglycerides) | 4 weeks
  Fasting blood samples will be collected to assess serum levels of total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL), Apo A (mg/dL), Apo B (mg/dL) and triglycerides (mg/dL) after 4 weeks of supplementation compared to baseline values.
Change from baseline in fasting blood glucose | 4 weeks
  Fasting blood glucose levels (mg/dl) will be measured at baseline and after 4 weeks of treatment to evaluate the effect of Berbevis™. Blood samples will be collected in the morning after at least 8 hours of fasting.
Change from baseline in fasting insulin | 4 weeks
  Fasting insulin levels (µIU/mL) will be assessed at baseline and after 4 weeks of treatment. Blood samples will be collected under fasting conditions to evaluate insulin secretion.
Change from baseline in HOMA-IR index | 4 weeks
  The Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) will be calculated using fasting glucose and insulin values at baseline and after 4 weeks of treatment to evaluate insulin resistance.
Change from baseline in glycated hemoglobin (HbA1c) | 4 weeks
  HbA1c levels (%) will be measured at baseline and after 4 weeks of treatment to evaluate longer-term glycemic control.
Change from baseline in C-reactive protein (CRP) | 4 weeks
  CRP levels (mg/L) will be evaluated at baseline and after 4 weeks of treatment to assess systemic inflammation.
Change from baseline in AST levels | 4 weeks
  AST serum levels (U/L) will be measured at baseline and after 4 weeks of treatment to assess liver function and potential hepatotoxicity.
Change from baseline in ALT levels | 4 weeks
  ALT serum levels (U/L) will be measured at baseline and after 4 weeks of treatment to evaluate liver cell integrity and potential hepatocellular damage.
Change from baseline in Gamma-GT levels | 4 weeks
  Gamma-GT levels (U/L) will be analyzed at baseline and after 4 weeks of treatment to monitor cholestasis or bile duct involvement.
Change from baseline in alkaline phosphatase levels | 4 weeks
  Alkaline phosphatase serum levels (U/L) will be measured at baseline and after 4 weeks of treatment to evaluate liver and bone metabolism.
Change from baseline in serum protein fractions (protein electrophoresis) | 4 weeks
  Serum protein fractions (e.g., albumin, alpha, beta, gamma globulins - g/dL) will be analyzed at baseline and after 4 weeks using protein electrophoresis to assess liver synthetic function and potential inflammation.
Change from baseline in lean mass and fat mass assessed by DEXA | 4 weeks
  Total body fat mass and whole-body lean mass (kg) will be measured using dual-energy X-ray absorptiometry (DEXA) at baseline and after 4 weeks to evaluate changes in fat-free body mass and body fat reduction or increase.
Change from baseline in visceral adipose tissue assessed by DEXA | From may 2025 to may 2026
  Visceral adipose tissue (cm²) will be estimated using DEXA at baseline and after 4 weeks to assess abdominal fat distribution and potential metabolic impact.

OTHER OUTCOMES:
Change from baseline in body weight | 4 weeks
  Body weight (kg) will be measured at baseline and after 4 weeks to evaluate potential weight changes due to the intervention.
Change from baseline in Body Mass Index (BMI) | 4 weeks
  BMI (kg/m²) will be calculated from weight and height measurements at baseline and after 4 weeks to assess changes in body composition.
Change from baseline in waist circumference | 4 weeks
  Waist circumference (cm) will be measured at baseline and after 4 weeks to evaluate changes in abdominal adiposity.